CLINICAL TRIAL: NCT05347381
Title: Selinexol Combined With Dexamethasone in the Treatment of CAEBV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Selinexor；Dexamethasone；CAEBV
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: CAEBV
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Selinexol and Dexamethasone (Experimental): Selinesol 20mg/tablet 60mg po qw first week, second week, biw third week, namely d1, d8, d15, d18.
  Dexamethasone 0.75mg/tablet 1.5mg po bid d1-21;
  Interventions: Drug: Selinexol and Dexamethasone

INTERVENTIONS:
Drug: Selinexol and Dexamethasone — Selinesol 20mg/tablet 60mg po qw first week, second week, biw third week, namely d1, d8, d15, d18.
  Dexamethasone 0.75mg/tablet 1.5mg po bid d1-21;

SUMMARY:
This study is a single-center, prospective, observational clinical study to evaluate the Effecive and Safty of Selinexol and Dexamethasone in CAEBV

ELIGIBILITY:
Inclusion Criteria:

-1) Age ≥14 years old, expected survival time is more than 3 months; 2) Any gender 3) CAEBV patients diagnosed by WHO criteria. 4) Eastern Cooperative Oncology Group (ECOG) physical status score of 0-1. 5) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) before the study ≤ 3 × upper limit of normal (ULN); total bilirubin ≤ 2 times the upper limit of normal; serum creatinine ≤ 1.5 times the normal value .

6) Absolute neutrophil count ≥1×109/L; platelets ≥50×109/L; hemoglobin ≥60 g/L. 7) International normalized ratio≤2.0, prothrombin time≤1.5×ULN. 8) Women of childbearing age must be confirmed by a pregnancy test that they are not pregnant, and are willing to take effective contraceptive measures during the trial and ≥ 12 months after the last dose; all male subjects during the study and ≥ 6 months after the last dose use of contraceptive methods; 9) The patients voluntarily joined the study, signed the informed consent, and had good compliance.

Exclusion Criteria:

* 1) There is evidence that EBV progresses to hemophagocytic syndrome; 2) Those who have participated in clinical trials of other drugs within 2 weeks; 3) Those with factors that affect oral drugs (such as inability to swallow, after gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.); 4) Those who have a history of psychotropic substance abuse and cannot quit or have mental disorders; 5) Uncontrolled infection (including lung infection, intestinal infection, etc.); active visceral hemorrhage (including gastrointestinal bleeding, alveolar hemorrhage, intracranial hemorrhage, etc.); and the investigators evaluate patients who will affect the safety of the trial.

  6) Cardiovascular disease of grade ≥2 (New York Heart Association Class 2 cardiovascular disease is defined as subjects who feel comfortable at rest but ordinary physical activity causes fatigue, palpitations, difficulty breathing or angina) 7) There is a significant medical history of renal, neurological, psychiatric, pulmonary, endocrine, metabolic, immune, and liver diseases, and the researcher believes that participating in this study will adversely affect him/her.

  8) Those who are known to be allergic to the study drug or its constituents.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
EBV-DNA | Change from before and 1,3,6 and 9 weeks after initiating Selinexol and Dexamethasone monotherapy
  Treatment effectiveness is defined: EBV-DNA copies/ml in peripheral blood turns negative, and the involved tissues (such as lymph nodes, bone marrow, skin, etc.) are negative in EBER test or the EBV copy number has decreased by more than 2 orders of magnitude, but it is still positive.
Progression Free Survival | 6 months
  rom date of inclusion to date of progression, relapse, or death from any cause
Adverse events | 6 months
  Adverse events including myelosuppression, infection, hemorrhage，vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China